CLINICAL TRIAL: NCT03392272
Title: Modified Müller's Muscle-conjunctival Resection Internal Ptosis Repair Using Fibrin Glue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Guy Ben-Simon, MD, Head, oculoplastic unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-17-4383-GBS
Record Dates: First submitted 2017-12-26; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Ptosis, Eyelid; Ptosis; Eyelid, Congenital; Surgical Procedure, Unspecified
Keywords: Ptosis; Müller's Muscle-Conjunctival Resection (MMCR); Fibrin Glue
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Intervention Model Description: A prospective randomized study
Who Masked: Care Provider
Masking Description: The physician will randomly assign the patient into the tisseel group or the sutures group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tisseel (Experimental): Müller's Muscle-Conjunctival Resection (MMCR) using glue instead of sutures
  Interventions: Device: Using of Tisseel fibrin glue
- Sutures (Active Comparator): Müller's Muscle-Conjunctival Resection (MMCR) using the usual procedure
  Interventions: Other: Using sutures

INTERVENTIONS:
Device: Using of Tisseel fibrin glue — Using of Tisseel fibrin glue instead of sutures in Müller's Muscle-Conjunctival Resection (MMCR) surgeries
  Arms: Tisseel
Other: Using sutures — Using sutures in Müller's Muscle-Conjunctival Resection (MMCR) surgeries
  Arms: Sutures

SUMMARY:
Fibrin glue is widely used in ophthalmology for homeostasis and tissue recovery. It is commonly used in ocular surface surgeries such as pterygium removal and conjunctival lesions excisions. In Müller's muscle-conjunctival resection (MMCR), sutures are used to reconnect the conjunctiva and Muller muscle, which causes discomfort and pain for the patient. The investigators' goal is to explore using fibrin glue instead of sutures in MMCR surgeries to shorten the procedure's length and alleviate patients discomfort and pain. This is especially important in the management of children suffering ptosis, where sedation and even general anaesthesia is required for sutured removal as a secondary procedure.

DETAILED DESCRIPTION:
Fibrin glue is widely used in ophthalmology for homeostasis and tissue recovery. It is commonly used in ocular surface surgeries such as pterygium removal and conjunctival lesions excisions.

Müller's muscle-conjunctival resection (MMCR) is the most common surgery for ptosis correction and is normally performed under local anaesthesia. In MMCR, a portion of the Muller and conjunctiva is resected, and sutures are used to reconnect the remaining edges. The suturing process requires several minutes and causes discomfort to the patient. In addition, many patients experience post operative discomfort due to the touch of the sutures in the superior ocular surface until their removal about 7-14 days post op. Moreover, the sutures removal process is commonly unpleasant, and in the pediatric patients requires sedation or general anaesthesia.

The investigators' goal is to explore using fibrin glue instead of sutures in MMCR surgeries to shorten the procedure's length and alleviate patients discomfort and pain. This is especially important in the management of children suffering ptosis, where sedation and even general anaesthesia is required for sutured removal as a secondary procedure.

Methods:

A prospective randomized study. Patients will be randomized into traditional MMCR using sutures, vs. MMCR using tisseel glue. Follow up will take place 1 day, 7 days, 1 month and 3 months post op. Main outcome measures included patient reported outcome such as pain grade and discomfort, and success of ptosis repair surgery defined by improvement in margin reflex distance, symmetry of upper eyelid position, and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

Patients with ptosis referred to Müller's Muscle-Conjunctival Resection (MMCR)

Exclusion Criteria:

Previous eyelid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain level | until 2 weeks post op
  Pain grade using visual analogue scale of 0-10 with 0=no pain and 10=worst pain.

SECONDARY OUTCOMES:
successful ptosis correction | 3 months
  satisfying improvement of margin to reflex distance

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Putterman AM, Urist MJ. Muller muscle-conjunctiva resection. Technique for treatment of blepharoptosis. Arch Ophthalmol. 1975 Aug;93(8):619-23. doi: 10.1001/archopht.1975.01010020595007. PMID 1156223
- [Background] Liu MT, Totonchi A, Katira K, Daggett J, Guyuron B. Outcomes of mild to moderate upper eyelid ptosis correction using Muller's muscle-conjunctival resection. Plast Reconstr Surg. 2012 Dec;130(6):799e-809e. doi: 10.1097/PRS.0b013e31826d9cb0. PMID 23190831
- [Background] Mercandetti M, Putterman AM, Cohen ME, Mirante JP, Cohen AJ. Internal levator advancement by Muller's muscle-conjunctival resection: technique and review. Arch Facial Plast Surg. 2001 Apr-Jun;3(2):104-10. doi: 10.1001/archfaci.3.2.104. PMID 11368662
- [Background] Carruth BP, Meyer DR. Simplified Muller's muscle-conjunctival resection internal ptosis repair. Ophthalmic Plast Reconstr Surg. 2013 Jan-Feb;29(1):11-4. doi: 10.1097/IOP.0b013e31826afb6b. PMID 23034694
- [Background] Zloto O, Greenbaum E, Fabian ID, Ben Simon GJ. Evicel versus Tisseel versus Sutures for Attaching Conjunctival Autograft in Pterygium Surgery: A Prospective Comparative Clinical Study. Ophthalmology. 2017 Jan;124(1):61-65. doi: 10.1016/j.ophtha.2016.09.010. Epub 2016 Nov 3. PMID 27817915